CLINICAL TRIAL: NCT02829307
Title: An Open Label Positron Emission Tomography (PET) Imaging Study Using 89Zirconium Labeled GSK3128349 to Investigate the Biodistribution and Clearance of an Albumin Binding Domain Antibody (AlbudAb) GSK3128349 Following Single Dose Intravenous Administration in Healthy Male Subjects
Brief Title: A Positron Emission Tomography (PET) Imaging Study to Investigate the Biodistribution and Clearance of an Albumin Binding Domain Antibody (AlbudAb) GSK3128349 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PRA Health Sciences for clinical study conduct. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 117169
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Results first posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-07

CONDITIONS: Drug-Related Side Effects and Adverse Reactions
Keywords: 89Zirconium; Open label; Pharmacokinetics; Radioactive; Clearance; Biodistribution
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 89Zr-GSK3128349 (Experimental): Subjects will receive a single dose of 89Zr-GSK3128349 as an intravenous (IV) infusion over 20 minutes to deliver a dose of 1 mg
  Interventions: Drug: 89Zr-GSK3128349 1 mg

INTERVENTIONS:
Drug: 89Zr-GSK3128349 1 mg — 89Zr-GSK3128349 is a mixture of unlabelled and zirconium-labelled GSK3128349, in the form of solution for IV administration, and is associated with about 15 MBq of radioactivity.

SUMMARY:
GSK3128349 is a small protein molecule (biopharmaceutical) that binds to albumin in the body, and by itself, has no pharmacological action. A pharmacologically active drug can be attached to GSK3128349 with the goal of changing the distribution and/or duration of action of the attached drug. This study will determine the distribution and pharmacokinetics (duration) of GSK3128349 itself after a single intravenous infusion. GSK3128349 has been labeled with and the radioisotope 89Zirconium allowing it to be visualized in the organs of the body using a PET scanner at multiple time points after GSK3128349 dosing. The data from this study will help predict the distribution of future drugs attached to GSK3128349. The total duration of a subject's participation is about approximately 10 weeks, including the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. - Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5x Upper Limit Normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Body Mass Index (BMI) within the range 19.0 - 31.0 kilogram (kg)/meter (m^2) (inclusive).
* Subjects must agree to use one of the contraception methods listed in the protocol.
* Capable of giving written informed consent, which includes compliance with the study requirements and restrictions.
* Average Corrected QT interval (QTc) <=450 milliseconds (msec)

Exclusion Criteria:

* Current evidence or history of an influenza-like illness.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of, or current, acute renal failure, known renal disease, or a renal disorder or abnormality that may compromise renal function. This includes having one kidney.
* Previous inclusion in a research and/or medical protocol involving nuclear medicine, PET or radiological investigations or occupational exposure that, together with the proposed study, will result in a total radiation exposure greater than 10 mSv over a 3 year period. Clinical exposure from which the subject receives a direct benefit (example, diagnostic test) is not included in these calculations.
* History of regular alcohol consumption within 6 months of the study defined as:

An average weekly intake of >21 units. One unit is equivalent to 8 g of alcohol: a half-pint (~240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.

* Unable to refrain from the use of prescription drugs within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study treatment, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Subject is a smoker >=5 cigarettes/day or with a smoking history of >5 pack years
* History of sensitivity to any of the study treatment or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Subject suffers from claustrophobia that limits the ability to remain still in the PET/CT scanner for the required amount of time.
* Subject has metal present in their body that will interfere with the PET/CT scanning.
* Estimate glomerular filtration rate (eGFR) <60 mL/min/1.73 m^2 (utilizing the Chronic Kidney Disease Epidemiology Collaboration (CKI-EPI) equation).
* Urine mg protein/mg creatinine Urine Protein Creatinine Ratio (UPCR) >0.3.
* Evidence of hematuria by urinalysis (1plus or greater dipstick test).
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C (Hep C) antibody result within 3 months of screening.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* A positive pre-study drug/alcohol screen.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Zuidlaren, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in Netherlands from 23-Aug-16 to 27-Jan-17. A total of 8 participants were randomized in the study who received 89Zr-GSK3128349 which was a mixture of unlabelled and zirconium-labelled GSK3128349, in the form of solution for intravenous (IV) administration.
Pre-assignment Details: A total of 34 participants were screened, of which 26 were screen failures. The reasons for screen failure were: did not meet the inclusion/exclusion criteria (11 participants) and investigator discretion (15 participants).
Groups:
- 89Zr-GSK3128349: Eligible participants received a single dose of 89Zr-GSK3128349 as an IV infusion over 20 minutes to deliver a dose of 1 milligram (mg).
Period: Overall Study
Arm/Group | 89Zr-GSK3128349
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Population comprised of all participants who received a dose of GSK3128349 radiolabelled with 89-zirconium (89Zr-GSK3128349).
Groups:
- 89Zr-GSK3128349: Eligible participants received a single dose of 89Zr-GSK3128349 as an IV infusion over 20 minutes to deliver a dose of 1 mg.
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.0 (2.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 1
  White- White/Caucasian/ European Heritage | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Standardized Uptake Values (SUVs) Derived From Positron Emission Tomography-Computer Tomography (PET-CT) Data
Description: SUV is a mathematically derived ratio of tissue radioactivity concentration and the injected dose of radioactivity per kilogram of the participant's body weight at a given point in time. SUV was analyzed for each region of interest (ROI) such as liver, kidney, muscle, spleen, heart, lung, bladder, thymus, and if feasible blood and bone. A maximum of 4 PET scans were conducted in each participant. Mean SUV derived from PET-CT has been presented.
Time Frame: Up to Day 7
Population: Pharmacokinetic (PK) Population comprised of participants in the Safety Population for whom a PK sample was obtained and analyzed, and/or for which a PET scan was completed. Only those participants available at the specified time points were analyzed represented by n=X in the category titles.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 8
Ratio
  Thigh muscle: PET scan 1; n=8 | 0.515 (0.1387)
  Thigh muscle: PET scan 2; n=8 | 0.566 (0.1315)
  Thigh muscle: PET scan 3; n=7: number analyzed (Participants) | 7
  Thigh muscle: PET scan 3; n=7 | 0.607 (0.0767)
  Thigh muscle: PET scan 4; n=7: number analyzed (Participants) | 7
  Thigh muscle: PET scan 4; n=7 | 0.623 (0.1509)
  Liver: PET scan 1; n=8 | 4.929 (0.7219)
  Liver: PET scan 2; n=8 | 3.231 (0.4981)
  Liver: PET scan 3; n=7: number analyzed (Participants) | 7
  Liver: PET scan 3; n=7 | 2.994 (0.7314)
  Liver: PET scan 4; n=7: number analyzed (Participants) | 7
  Liver: PET scan 4; n=7 | 2.280 (0.3151)
  Pancreas: PET scan 1; n=7: number analyzed (Participants) | 7
  Pancreas: PET scan 1; n=7 | 2.177 (0.4573)
  Pancreas: PET scan 2; n=7: number analyzed (Participants) | 7
  Pancreas: PET scan 2; n=7 | 2.029 (0.6621)
  Pancreas: PET scan 3; n=6: number analyzed (Participants) | 6
  Pancreas: PET scan 3; n=6 | 1.887 (0.4131)
  Pancreas: PET scan 4; n=6: number analyzed (Participants) | 6
  Pancreas: PET scan 4; n=6 | 1.917 (1.0314)
  Thyroid gland: PET scan 1; n=8 | 2.338 (0.8821)
  Thyroid gland: PET scan 2; n=8 | 2.171 (0.8408)
  Thyroid gland: PET scan 3; n=7: number analyzed (Participants) | 7
  Thyroid gland: PET scan 3; n=7 | 2.330 (1.0510)
  Thyroid gland: PET scan 4; n=7: number analyzed (Participants) | 7
  Thyroid gland: PET scan 4; n=7 | 1.789 (0.4791)
  Testis: PET scan 1; n=8 | 3.336 (0.7479)
  Testis: PET scan 2; n=8 | 3.733 (0.7793)
  Testis: PET scan 3; n=7: number analyzed (Participants) | 7
  Testis: PET scan 3; n=7 | 3.259 (0.9988)
  Testis: PET scan 4; n=7: number analyzed (Participants) | 7
  Testis: PET scan 4; n=7 | 3.280 (0.4789)
  Bladder: PET scan 1; n=8 | 2.750 (1.0483)
  Bladder: PET scan 2; n=8 | 1.149 (0.4572)
  Bladder: PET scan 3; n=7: number analyzed (Participants) | 7
  Bladder: PET scan 3; n=7 | 1.630 (0.4938)
  Bladder: PET scan 4; n=7: number analyzed (Participants) | 7
  Bladder: PET scan 4; n=7 | 1.609 (0.4176)
  Kidney: PET scan 1; n=8 | 7.845 (1.1487)
  Kidney: PET scan 2; n=8 | 9.516 (1.0005)
  Kidney: PET scan 3; n=7: number analyzed (Participants) | 7
  Kidney: PET scan 3; n=7 | 10.466 (2.2765)
  Kidney: PET scan 4; n=7: number analyzed (Participants) | 7
  Kidney: PET scan 4; n=7 | 8.603 (1.6626)
  Parotid gland: PET scan 1; n=8 | 1.514 (0.3005)
  Parotid gland: PET scan 2; n=8 | 1.430 (0.3091)
  Parotid gland: PET scan 3; n=7: number analyzed (Participants) | 7
  Parotid gland: PET scan 3; n=7 | 1.541 (0.2084)
  Parotid gland: PET scan 4; n=7: number analyzed (Participants) | 7
  Parotid gland: PET scan 4; n=7 | 1.531 (0.1643)
  Bone marrow: PET scan 1; n=8 | 1.746 (0.2575)
  Bone marrow: PET scan 2; n=8 | 1.378 (0.2066)
  Bone marrow: PET scan 3; n=7: number analyzed (Participants) | 7
  Bone marrow: PET scan 3; n=7 | 1.289 (0.2998)
  Bone marrow: PET scan 4; n=7: number analyzed (Participants) | 7
  Bone marrow: PET scan 4; n=7 | 1.350 (0.2802)
  Spleen: PET scan 1; n=8 | 5.220 (0.6398)
  Spleen: PET scan 2; n=8 | 3.691 (0.4638)
  Spleen: PET scan 3; n=7: number analyzed (Participants) | 7
  Spleen: PET scan 3; n=7 | 3.296 (0.8611)
  Spleen: PET scan 4; n=7: number analyzed (Participants) | 7
  Spleen: PET scan 4; n=7 | 3.097 (0.4946)
  Brain: PET scan 1; n=8 | 0.461 (0.0762)
  Brain: PET scan 2; n=8 | 0.295 (0.0901)
  Brain: PET scan 3; n=7: number analyzed (Participants) | 7
  Brain: PET scan 3; n=7 | 0.231 (0.0689)
  Brain: PET scan 4; n=7: number analyzed (Participants) | 7
  Brain: PET scan 4; n=7 | 0.201 (0.0348)
  Lung: PET scan 1; n=8 | 1.884 (0.5968)
  Lung: PET scan 2; n=8 | 1.345 (0.4381)
  Lung: PET scan 3; n=7: number analyzed (Participants) | 7
  Lung: PET scan 3; n=7 | 1.186 (0.4720)
  Lung: PET scan 4; n=7: number analyzed (Participants) | 7
  Lung: PET scan 4; n=7 | 0.893 (0.2583)
  Aorta: PET scan 1; n=8 | 10.835 (2.0289)
  Aorta: PET scan 2; n=8 | 6.573 (1.5621)
  Aorta: PET scan 3; n=7: number analyzed (Participants) | 7
  Aorta: PET scan 3; n=7 | 5.516 (1.4879)
  Aorta: PET scan 4; n=7: number analyzed (Participants) | 7
  Aorta: PET scan 4; n=7 | 4.299 (0.8195)
  Heart: PET scan 1; n=8 | 8.601 (1.8566)
  Heart: PET scan 2; n=8 | 5.851 (1.5742)
  Heart: PET scan 3; n=7: number analyzed (Participants) | 7
  Heart: PET scan 3; n=7 | 4.829 (1.3661)
  Heart: PET scan 4; n=7: number analyzed (Participants) | 7
  Heart: PET scan 4; n=7 | 3.701 (0.6770)
  Kidney, cortex: PET scan 1; n=8 | 8.805 (1.4835)
  Kidney, cortex: PET scan 2; n=8 | 12.145 (1.7704)
  Kidney, cortex: PET scan 3; n=7: number analyzed (Participants) | 7
  Kidney, cortex: PET scan 3; n=7 | 11.966 (1.5492)
  Kidney, cortex: PET scan 4; n=7: number analyzed (Participants) | 7
  Kidney, cortex: PET scan 4; n=7 | 10.479 (1.6047)
  Kidney, medulla: PET scan 1; n=8 | 6.996 (1.5577)
  Kidney, medulla: PET scan 2; n=8 | 7.416 (1.2101)
  Kidney, medulla: PET scan 3; n=7: number analyzed (Participants) | 7
  Kidney, medulla: PET scan 3; n=7 | 8.247 (2.3436)
  Kidney, medulla: PET scan 4; n=7: number analyzed (Participants) | 7
  Kidney, medulla: PET scan 4; n=7 | 6.691 (1.1767)
  Body: PET scan 1; n=8 | 0.739 (0.1647)
  Body: PET scan 2; n=8 | 0.654 (0.1632)
  Body: PET scan 3; n=7: number analyzed (Participants) | 7
  Body: PET scan 3; n=7 | 0.701 (0.1728)
  Body: PET scan 4; n=7: number analyzed (Participants) | 7
  Body: PET scan 4; n=7 | 0.631 (0.1680)

2. Primary Outcome: Mean Volume of ROI for Each Organ at All Time Points
Description: Volume of ROI is the volume specified in organs as measured in PET or CT images. Mean volume of ROI for each organ has been presented.
Time Frame: Up to Day 7
Population: PK Population. Only those participants available at the specified time points were analyzed represented by n=X in the category titles.
Measure: Mean (Standard Deviation); unit: Milliliter (mL)
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 8
Milliliter (mL)
  Thigh muscle: PET scan 1; n=8 | 45.001 (16.6069)
  Thigh muscle: PET scan 2; n=8 | 40.975 (12.4102)
  Thigh muscle: PET scan 3; n=7: number analyzed (Participants) | 7
  Thigh muscle: PET scan 3; n=7 | 40.094 (6.7137)
  Thigh muscle: PET scan 4; n=7: number analyzed (Participants) | 7
  Thigh muscle: PET scan 4; n=7 | 38.874 (10.7444)
  Liver: PET scan 1; n=8 | 574.546 (301.4580)
  Liver: PET scan 2; n=8 | 532.373 (147.3186)
  Liver: PET scan 3; n=7: number analyzed (Participants) | 7
  Liver: PET scan 3; n=7 | 488.974 (156.2512)
  Liver: PET scan 4; n=7: number analyzed (Participants) | 7
  Liver: PET scan 4; n=7 | 496.861 (166.0174)
  Pancreas: PET scan 1; n=7: number analyzed (Participants) | 7
  Pancreas: PET scan 1; n=7 | 7.777 (3.3295)
  Pancreas: PET scan 2; n=7: number analyzed (Participants) | 7
  Pancreas: PET scan 2; n=7 | 7.780 (2.7156)
  Pancreas: PET scan 3; n=6: number analyzed (Participants) | 6
  Pancreas: PET scan 3; n=6 | 5.905 (3.0366)
  Pancreas: PET scan 4; n=6: number analyzed (Participants) | 6
  Pancreas: PET scan 4; n=6 | 6.877 (4.7283)
  Thyroid gland: PET scan 1; n=8 | 2.750 (1.5549)
  Thyroid gland: PET scan 2; n=8 | 3.004 (0.9845)
  Thyroid gland: PET scan 3; n=7: number analyzed (Participants) | 7
  Thyroid gland: PET scan 3; n=7 | 2.913 (0.9590)
  Thyroid gland: PET scan 4; n=7: number analyzed (Participants) | 7
  Thyroid gland: PET scan 4; n=7 | 4.137 (2.0853)
  Testis: PET scan 1; n=8 | 13.223 (6.7226)
  Testis: PET scan 2; n=8 | 12.010 (6.5955)
  Testis: PET scan 3; n=7: number analyzed (Participants) | 7
  Testis: PET scan 3; n=7 | 11.583 (4.5054)
  Testis: PET scan 4; n=7: number analyzed (Participants) | 7
  Testis: PET scan 4; n=7 | 13.871 (7.6413)
  Bladder: PET scan 1; n=8 | 84.228 (69.2024)
  Bladder: PET scan 2; n=8 | 60.669 (26.7843)
  Bladder: PET scan 3; n=7: number analyzed (Participants) | 7
  Bladder: PET scan 3; n=7 | 54.771 (26.2373)
  Bladder: PET scan 4; n=7: number analyzed (Participants) | 7
  Bladder: PET scan 4; n=7 | 66.291 (47.1061)
  Kidney: PET scan 1; n=8 | 144.093 (32.8834)
  Kidney: PET scan 2; n=8 | 162.578 (55.1273)
  Kidney: PET scan 3; n=7: number analyzed (Participants) | 7
  Kidney: PET scan 3; n=7 | 152.031 (36.5278)
  Kidney: PET scan 4; n=7: number analyzed (Participants) | 7
  Kidney: PET scan 4; n=7 | 177.840 (30.9614)
  Parotid gland: PET scan 1; n=8 | 8.304 (3.5772)
  Parotid gland: PET scan 2; n=8 | 9.391 (4.2224)
  Parotid gland: PET scan 3; n=7: number analyzed (Participants) | 7
  Parotid gland: PET scan 3; n=7 | 8.611 (1.6606)
  Parotid gland: PET scan 4; n=7: number analyzed (Participants) | 7
  Parotid gland: PET scan 4; n=7 | 9.896 (2.6622)
  Bone marrow: PET scan 1; n=8 | 36.625 (18.3824)
  Bone marrow: PET scan 2; n=8 | 37.495 (15.1968)
  Bone marrow: PET scan 3; n=7: number analyzed (Participants) | 7
  Bone marrow: PET scan 3; n=7 | 45.271 (18.2245)
  Bone marrow: PET scan 4; n=7: number analyzed (Participants) | 7
  Bone marrow: PET scan 4; n=7 | 42.871 (14.4365)
  Spleen: PET scan 1; n=8 | 62.238 (20.6549)
  Spleen: PET scan 2; n=8 | 67.160 (21.9034)
  Spleen: PET scan 3; n=7: number analyzed (Participants) | 7
  Spleen: PET scan 3; n=7 | 54.544 (13.4153)
  Spleen: PET scan 4; n=7: number analyzed (Participants) | 7
  Spleen: PET scan 4; n=7 | 47.474 (18.3678)
  Brain: PET scan 1; n=8 | 575.996 (91.2147)
  Brain: PET scan 2; n=8 | 510.614 (139.8124)
  Brain: PET scan 3; n=7: number analyzed (Participants) | 7
  Brain: PET scan 3; n=7 | 471.550 (152.8605)
  Brain: PET scan 4; n=7: number analyzed (Participants) | 7
  Brain: PET scan 4; n=7 | 498.207 (145.5429)
  Lung: PET scan 1; n=8 | 329.891 (134.1686)
  Lung: PET scan 2; n=8 | 329.374 (162.8302)
  Lung: PET scan 3; n=7: number analyzed (Participants) | 7
  Lung: PET scan 3; n=7 | 328.794 (115.2736)
  Lung: PET scan 4; n=7: number analyzed (Participants) | 7
  Lung: PET scan 4; n=7 | 308.494 (77.7344)
  Aorta: PET scan 1; n=8 | 6.388 (2.9532)
  Aorta: PET scan 2; n=8 | 8.171 (3.5471)
  Aorta: PET scan 3; n=7: number analyzed (Participants) | 7
  Aorta: PET scan 3; n=7 | 7.887 (3.1780)
  Aorta: PET scan 4; n=7: number analyzed (Participants) | 7
  Aorta: PET scan 4; n=7 | 8.199 (3.5405)
  Heart: PET scan 1; n=8 | 135.013 (74.5105)
  Heart: PET scan 2; n=8 | 111.133 (53.4101)
  Heart: PET scan 3; n=7: number analyzed (Participants) | 7
  Heart: PET scan 3; n=7 | 105.007 (26.1510)
  Heart: PET scan 4; n=7: number analyzed (Participants) | 7
  Heart: PET scan 4; n=7 | 103.971 (40.0218)
  Kidney, cortex: PET scan 1; n=8 | 5.483 (3.0342)
  Kidney, cortex: PET scan 2; n=8 | 5.728 (2.7257)
  Kidney, cortex: PET scan 3; n=7: number analyzed (Participants) | 7
  Kidney, cortex: PET scan 3; n=7 | 6.770 (1.2609)
  Kidney, cortex: PET scan 4; n=7: number analyzed (Participants) | 7
  Kidney, cortex: PET scan 4; n=7 | 7.229 (3.5309)
  Kidney, medulla: PET scan 1; n=8 | 4.646 (2.1984)
  Kidney, medulla: PET scan 2; n=8 | 4.885 (2.3112)
  Kidney, medulla: PET scan 3; n=7: number analyzed (Participants) | 7
  Kidney, medulla: PET scan 3; n=7 | 6.104 (1.4927)
  Kidney, medulla: PET scan 4; n=7: number analyzed (Participants) | 7
  Kidney, medulla: PET scan 4; n=7 | 6.661 (3.3183)
  Body: PET scan 1; n=8 | 103654.675 (29591.9710)
  Body: PET scan 2; n=8 | 106925.973 (32398.3328)
  Body: PET scan 3; n=7: number analyzed (Participants) | 7
  Body: PET scan 3; n=7 | 96034.243 (22195.6206)
  Body: PET scan 4; n=7: number analyzed (Participants) | 7
  Body: PET scan 4; n=7 | 100291.249 (27671.1649)

3. Secondary Outcome: Area Under Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (AUC [0-t]) and Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinite Time (AUC [0-inf]) of 89Zr-GSK3128349 and GSK3128349
Description: PK parameters included AUC (0-t) and AUC (0-inf). AUC (0-t) and AUC (0-inf) for 89Zr-GSK3128349 was calculated from the whole blood and plasma concentration-time data, measured by scintillation counting. AUC (0-t) and AUC (0-inf) for GSK3128349 was calculated from the whole blood and plasma concentration-time data, measured by mass spectrometry.
Time Frame: Pre-dose, 1 hour (h), 3 h, 6 h, 8h, 24 h post-dose, Day 4, Day 6, Day 14, Day 22, Day 33 and Day 45
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (Becquerel [Bq] per mL)*h
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 7
(Becquerel [Bq] per mL)*h
  89Zr-GSK3128349: AUC (0-t) | 461526.5722 (11.1647)
  89Zr-GSK3128349: AUC (0-inf) | 930260.1961 (19.4399)
  GSK3128349: AUC (0-t) | 82177.6360 (19.0961)
  GSK3128349: AUC (0-inf) | 104257.7700 (16.5839)

4. Secondary Outcome: Percent Area Under the Curve Obtained by Extrapolation (AUCex) and Percent Area Under the First Moment Curve Obtained by Extrapolation (AUMCex) of 89Zr-GSK3128349 and GSK3128349
Description: PK parameters included AUCex and AUMCex. AUCex and AUMCex for 89Zr-GSK3128349 was calculated from the whole blood and plasma concentration-time data, measured by scintillation counting. AUCex and AUMCex for GSK3128349 was calculated from the whole blood and plasma concentration-time data, measured by mass spectrometry.
Time Frame: Pre-dose, 1 h, 3 h, 6 h, 8h, 24 h post-dose, Day 4, Day 6, Day 14, Day 22, Day 33 and Day 45
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage area under the curve
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 7
Percentage area under the curve
  89Zr-GSK3128349: Percent AUCex | 48.5838 (20.4243)
  89Zr-GSK3128349: Percent AUMCex | 84.0346 (8.3187)
  GSK3128349: Percent AUCex | 20.7353 (19.8191)
  GSK3128349: Percent AUMCex | 55.9698 (11.6540)

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of 89Zr-GSK3128349
Description: PK parameters included Cmax. Cmax for 89Zr-GSK3128349 was calculated from the whole blood and plasma concentration-time data, measured by scintillation counting.
Time Frame: Pre-dose, 1 h, 3 h, 6 h, 8h, 24 h post-dose, Day 4, Day 6, Day 14, Day 22, Day 33 and Day 45
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Bq per mL
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 7
Bq per mL | 3872.7027 (8.6104)

6. Secondary Outcome: Cmax of GSK3128349
Description: PK parameters included Cmax. Cmax for GSK3128349 was calculated from the whole blood and plasma concentration-time data, measured by mass spectrometry.
Time Frame: Pre-dose, 1 h, 3 h, 6 h, 8h, 24 h post-dose, Day 4, Day 6, Day 14, Day 22, Day 33 and Day 45
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram (ng) per mL
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 7
Nanogram (ng) per mL | 374.3868 (10.4183)

7. Secondary Outcome: Apparent Terminal Phase Half-life (t1/2) and Mean Residence Time (MRT) of 89Zr-GSK3128349 and GSK3128349
Description: PK parameters included t1/2 and MRT. t1/2 and MRT for 89Zr-GSK3128349 was calculated from the whole blood and plasma concentration-time data, measured by scintillation counting. t1/2 and MRT for GSK3128349 was calculated from the whole blood and plasma concentration-time data, measured by mass spectrometry.
Time Frame: Pre-dose, 1 h, 3 h, 6 h, 8h, 24 h post-dose, Day 4, Day 6, Day 14, Day 22, Day 33 and Day 45
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 7
Hours
  89Zr-GSK3128349: t1/2 | 279.3697 (40.6517)
  89Zr-GSK3128349: MRT | 404.8882 (36.4904)
  GSK3128349: t1/2 | 420.6105 (9.2835)
  GSK3128349: MRT | 562.3356 (9.7841)

8. Secondary Outcome: Elimination Rate Constant (Lambda-z) of 89Zr-GSK3128349
Description: PK parameters included lambda-z. Cmax for 89Zr-GSK3128349 was calculated from the whole blood and plasma concentration-time data, measured by scintillation counting.
Time Frame: Pre-dose, 1 h, 3 h, 6 h, 8h, 24 h post-dose, Day 4, Day 6, Day 14, Day 22, Day 33 and Day 45
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1 per h
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 7
1 per h | 0.0025 (40.6517)

9. Secondary Outcome: Volume of Distribution at a Steady State (Vss) and Volume of Distribution in the Terminal Phase (Vz) of 89Zr-GSK3128349 and GSK3128349
Description: PK parameters included Vss and Vz. Vss and Vz for 89Zr-GSK3128349 was calculated from the whole blood and plasma concentration-time data, measured by scintillation counting. Vss and Vz for GSK3128349 was calculated from the whole blood and plasma concentration-time data, measured by mass spectrometry.
Time Frame: Pre-dose, 1 h, 3 h, 6 h, 8h, 24 h post-dose, Day 4, Day 6, Day 14, Day 22, Day 33 and Day 45
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 7
mL
  89Zr-GSK3128349: Vss | 5440.5241 (21.7532)
  89Zr-GSK3128349: Vz | 5415.7602 (25.5996)
  GSK3128349: Vss | 5393.6763 (13.5175)
  GSK3128349: Vz | 5820.3069 (13.9190)

10. Secondary Outcome: Area Under the First Moment Curve From Pre-dose Extrapolated to Infinite Time (AUMC [0-inf]) and Area Under the First Moment Curve From Pre-dose Extrapolated to Last Time of Quantifiable Concentration (AUMC [0-t]) of 89Zr-GSK3128349
Description: PK parameters included AUMC (0-inf) and AUMC (0-t). AUMC (0-inf) and AUMC (0-t) for 89Zr-GSK3128349 was calculated from the whole blood and plasma concentration-time data, measured by scintillation counting.
Time Frame: Pre-dose, 1 h, 3 h, 6 h, 8h, 24 h post-dose, Day 4, Day 6, Day 14, Day 22, Day 33 and Day 45
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (Bq/mL)*h^2)
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 7
(Bq/mL)*h^2)
  89Zr-GSK3128349: AUMC (0-inf) | 376651413.6839 (56.6074)
  89Zr-GSK3128349: AUMC (0-t) | 53242134.4377 (10.0977)

11. Secondary Outcome: AUMC (0-inf) and AUMC (0-t) of GSK3128349
Description: PK parameters included AUMC (0-inf) and AUMC (0-t). AUMC (0-inf) and AUMC (0-t) for GSK3128349 was calculated from the whole blood and plasma concentration-time data, measured by mass spectrometry.
Time Frame: Pre-dose, 1 h, 3 h, 6 h, 8h, 24 h post-dose, Day 4, Day 6, Day 14, Day 22, Day 33 and Day 45
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng/mL)*h^2
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 7
(ng/mL)*h^2
  GSK3128349: AUMC (0-inf) | 58627561.8533 (23.8246)
  GSK3128349: AUMC (0-t) | 25366300.3864 (31.7095)

12. Secondary Outcome: Clearance of 89Zr-GSK3128349 and GSK3128349
Description: PK parameters included clearance. Clearance for 89Zr-GSK3128349 was calculated from the whole blood and plasma concentration-time data, measured by scintillation counting. Clearance for GSK3128349 was calculated from the whole blood and plasma concentration-time data, measured by mass spectrometry.
Time Frame: Pre-dose, 1 h, 3 h, 6 h, 8h, 24 h post-dose, Day 4, Day 6, Day 14, Day 22, Day 33 and Day 45
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 7
mL/h
  89Zr-GSK3128349: Clearance | 13.4371 (19.4399)
  GSK3128349: Clearance | 9.5918 (16.5657)

13. Secondary Outcome: Mean Organ and Effective Dose
Description: Organ dose was defined as the amount of radiation delivered to a particular organ. Effective dose was defined as the tissue-weighted sum of the organ doses in all specified tissues and organs of the human body. The organ and effective dose is a fraction of milliSievert (mSv) and MegaBecquerel (MBq). The mean relative uptake of 89Zr-GSK3128349 in different organs for all participants across all PET scans is presented.
Time Frame: Up to Day 7
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mSv/MBq
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 7
mSv/MBq
  Liver | 0.7909 (0.15549)
  Pancreas | 0.5701 (0.09391)
  Thyroid gland | 0.4004 (0.09722)
  Testis | 0.4827 (0.03345)
  Bladder | 0.2889 (0.02315)
  Kidney | 1.3871 (0.30625)
  Bone marrow | 0.3407 (0.03146)
  Spleen | 0.7314 (0.08562)
  Thymus gland | 0.3457 (0.03229)
  Brain | 0.1431 (0.04001)
  Lung | 0.8413 (0.17595)
  Heart | 0.6721 (0.14849)
  Body | 0.4480 (0.03811)

14. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant or is associated with liver injury or impaired liver function.
Time Frame: Up to 45 days
Population: Safety Population which comprised of all participants who received a dose of 89Zr-GSK3128349.
Measure: Number; unit: Participants
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 8
Participants
  AE | 2
  SAE | 0

15. Secondary Outcome: Number of Participants With Clinical Chemistry Data of Potential Clinical Concern
Description: The potential clinical concern range for clinical chemistry parameters were: glucose (low: < 3 millimole [mmol]/L and high: > 9 mmol/L), creatinine (high: Change from Baseline or Day 1 should be positive and > 44.2 mmol/L), phosphorous (low: < 0.8 mmol/L and high: > 1.6 mmol/L), magnesium (low: < 0.5 mmol/L and high: > 1.23 mmol/L), calcium (low: <2 mmoL/L and high: > 2.75 mmol/L), carbon dioxide content (low: < 18 mmol/L and high: > 32 mmol/L), albumin (low: < 30 mmol/L), potassium (low: < 3.0 mmol/L and high: > 5.5 mmol/L) and sodium (low: < 130 mmol/L and high: > 130 mmol/L). Number of participants with clinical chemistry abnormalities of potential clinical importance are presented
Time Frame: Up to 45 days
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 8
Participants | 0

16. Secondary Outcome: Number of Participants With Hematology Data of Potential Clinical Concern
Description: The potential clinical concern range for hematology parameters were: Hemoglobin (low: > 25 gram per Liter change from Baseline/Day 1 and high: > 180 gram per Liter), lymphocytes (low: < 0.8 gigacells/L), hematocrit (low: > 0.075 ratio change from Baseline and high: > 0.54 ratio), neutrophil count (low: < 1.5*10^9/Liter), platelet count (low: < 100 gigacells/L and high: > 550 gigacells/L), white blood cell (WBC) count (low: < 3 gigacells/L and high: > 20 gigacells/L). Number of participants with hematology abnormalities of potential clinical importance are presented.
Time Frame: Up to 45 days
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 8
Participants | 0

17. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Values of Potential Clinical Concern
Description: ECG measurements were made with the participant in a supine position having rested in this position for at least 5 minutes before each reading. Triplicate 12-lead ECGS were obtained pre dose at Day 1 and single 12-lead ECGs will be obtained at other time points during the study. The potential clinical concern range for ECG parameters was as follows: Absolute corrected QT (QTc) interval (lower: >450 milliseconds [msec], >450 msec, >=480 msec and >=500 msec) and (higher: <=479 msec and <=499 msec); absolute PR interval (lower: <110 and higher >220 msec) and absolute QRS interval (lower: <75 msec and >110 msec). Number of participants with ECG values of potential clinical concern are presented.
Time Frame: Pre-dose on Day 1, 1 h and 24 h post-dose on Day 1 and Day 45
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 8
Participants
  QRS duration | 1
  Heart rate | 0
  PR interval | 0
  RR interval | 0
  QT interval | 0
  QT interval corrected by Bazett's formula | 0
  QT interval corrected by Fridericia formula | 0

18. Secondary Outcome: Number of Participants With Vital Signs of Potential Clinical Concern
Description: Vital signs included pulse rate, systolic and diastolic blood pressure and body temperature. All vital sign measurements were made with the participant in a supine position and rested in this position for at least 5 minutes before each reading. The potential clinical concern range for systolic blood pressure: <85 and >160 millimeters of mercury (mmHg), for diastolic: <45 and >100 mmHg and heart rate: <40 and >110 beats per minute. Number of participants with vital signs of potential clinical concern are presented.
Time Frame: Up to 45 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 8
Participants | 0

19. Secondary Outcome: Number of Participants With Positive Anti-GSK3128349 Antibody Assay
Description: Blood samples for testing antibodies against GSK3128349 will be collected on Day 1 (pre-dose) and on Day 43. The actual date and time of each blood sample collection was recorded. The first blood sample was taken pre-dose on Day 1 to determine the presence, if any, of pre-existing Anti Drug Antibodies (ADAs). The presence of such antibodies was assessed using an electrochemiluminescent (ECL) immuno assay. If sera contain anti-GSK3128349 antibodies, they were further analyzed for the antibody specificity and titres. Number of participants who were found to have anti-GSK3128349 antibodies are presented.
Time Frame: Pre-dose on Day 1 and Day 43
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 8
Participants | 1

20. Secondary Outcome: Serum Titers of Anti-GSK3128349 Antibodies
Description: Blood samples for testing antibodies against GSK3128349 will be collected on Day 1 (pre-dose) and on Day 43. The actual date and time of each blood sample collection was recorded. The first blood sample was taken pre-dose on Day 1 to determine the presence, if any, of pre-existing ADAs. The presence of such antibodies and serum titers of anti-GSK3128349 antibodies was assessed using an ECL immuno-assay. If sera contain anti-GSK3128349 antibodies, they were further analyzed for the antibody specificity and titers.
Time Frame: Pre-dose on Day 1 and Day 43
Population: Safety Population. Only those participants with positive anti-GSK3128349 antibody assay were analyzed.
Measure: Mean (Standard Deviation); unit: Titers
Arm/Group | 89Zr-GSK3128349
Number analyzed (Participants) | 1
Titers
  Day 1, pre-dose | 80 (NA) — NA indicates Not Available because single participant was analyzed so Standard deviation could not be derived.
  Day 43 | 40 (NA) — NA indicates Not Available because single participant was analyzed so Standard deviation could not be derived.

ADVERSE EVENTS:
Time Frame: Up to 45 days
Description: SAE and non-SAE are reported for the Safety Population which comprised of all participants who received a dose of 89Zr-GSK3128349.
Arm/Group | 89Zr-GSK3128349
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 89Zr-GSK3128349 (N=8)
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Flatulence (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-05-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT02829307/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT02829307/SAP_001.pdf